CLINICAL TRIAL: NCT01897272
Title: Post-Operative Splinting After Short-Incision Carpal Tunnel Release: a Prospective, Randomized Study
Brief Title: Post-Operative Splinting After Short-Incision Carpal Tunnel Release: a Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Christine M. Kleinert Institute for Hand and Microsurgery (Other)
Responsible Party: Sponsor
Other Study IDs: 12.0416
Record Dates: First submitted 2013-06-13; First posted 2013-07-11 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; splinting; nerve decompression
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Splints

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Splinting After Surgery: This group will be fitted for a splint and given instructions on wearing their splint after their short-incision Carpal Tunnel Release
  Interventions: Behavioral: Splinting
- No Splinting After Surgery: This group will not be splinted after the short-incision carpal tunnel release

INTERVENTIONS:
Behavioral: Splinting — One group will have their wrist splinted after their carpal tunnel release surgery.
  Groups: Splinting After Surgery

SUMMARY:
This research study is for patients who are schedule to have carpal tunnel release surgery. The investigators have developed this study in order to determine if post-operative splinting is effective in improvement of patient outcomes after this surgical procedure. The study is being conducted under the direction of Huey Tien, MD. The purpose of this study is to determine if post-operative splinting is effective in improving patient outcomes after having short-incision carpal tunnel release. The investigators will randomize each patient into group 1, splinting after surgery or group 2 no splinting after surgery. Each group will have the same outcome measurements done to determine the best outcome of the two groups.

DETAILED DESCRIPTION:
Your participation in this study will last for five office visits of approximately 30 minutes each. If you decide to participate in this study, we would first have you come to clinic where you would undergo some standard measurements. This includes measuring grip and key pinch strength and completing a patient questionnaire. During your visits we will scan the cross-sectional area of the median nerve at the pisiform bone level to determine the level of CTS with the Ultrasound Biomiscroscopy machine (Vevo 2100). This is a new technique with a machine similar to a regular ultrasound machine. The primary difference is that the frequency of soundwaves is higher than a standard ultrasound machine. There are no known significant risks associated with the use of this machine. At this time the machine is experimental, and is not currently approved by the FDA for clinical use. However, this device is not considered to pose significant risk. Candidates for this study must have been diagnosed with single carpal tunnel syndrome and are going to receive nerve decompression with short incision, over the age of 18, and able to give informed consent to participate in a research study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with carpal tunnel syndrome and are going to receive nerve decompression with short incision
* The Criteria of CTS
* Numbness, tingling, pain and night symptoms in median nerve distribution
* Positive Tinel signs over the median nerve at the Carpal Tunnel
* Negative Tinel signs at the Supraclavicular and Infraclavicular areas
* Positive Carpal Tunnel Tests
* Electrophysiological changes (confirmed with NCT)
* Over the age of 18
* Ability to give informed consent to participate in a research study

Exclusion Criteria:

* Patients with peripheral neuropathy of the median nerve secondary to trauma, external compressions (tumours, bone malunion) or other non-compressive causes.
* Patients with the presence of Thoracic Outlet Syndrome (Tinel must be negative at the Supraclavicular and Infraclavicular areas)
* Patients with the presence of Cervical Disc disease
* Patients with another site of compression (such as pronator teres compression)
* Patients who have had previous carpal tunnel release on the same hand
* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We are looking for patients who are old enough to give informed consent who are preparing to have nerve decompression with short incision for their carpal tunnel syndrome.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Biomicroscopy of the cross section area of the median nerve at the pisiform level | Up to two years
  This is a high resolution ultrasound used to determine the distance between the surface and the median nerve. This device is a research device not approved for clinical use, but is considered a non-significant risk (NSR) device. This machine is just like a regular ultrasound machine. The primary difference is that the frequence of the soundwaves is higher than a standard ultrasound machine. At this time, the machine is experimental, and it is not currently approved by the FDA for clinical use. However, this same technology is used in similar devices by opthamologists to image retinas. It has been used on hudnreds of humans for research studies.

SECONDARY OUTCOMES:
Key Pinch Strength | Up to two years
Grip Strength | Up to two years
DASH questionnaire | Up to two years

CONTACTS AND LOCATIONS:
Overall Officials: Huey Tien, MD, Principal Investigator — Christine M. Kleinert Institute for Hand and Microsurgery; Millicent L Horn, BS, Study Chair — Christine M. Kleinert Institute for Hand and Microsurgery
Locations (2):
- United States (2):
  - Christine M. Kleinert Institute for Hand and Microsurgery, Louisville, Kentucky
  - Kleinert, Kutz & Associates, Louisville, Kentucky